CLINICAL TRIAL: NCT03477565
Title: Effectiveness of Kinesio Tex Tape Application in Reducing Edema and Seroma Formation Following Complex Reconstructive Breast Surgery
Brief Title: Kinesio Tex Tape in Reducing Edema and Seroma After Complex Reconstructive Breast Surgery
Acronym: BREASTAPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Stefano Martella, Primary Doctor of General Reconstructive Surgery Operating Unit., IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TAP_Sett17
Record Dates: First submitted 2018-02-17; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer; Mastectomy; Breast Implantation; Edema; Seroma
MeSH Terms: conditions — Breast Neoplasms; Edema; Seroma | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sperimental group (Experimental): Patients who belong to the sperimental group ("SPER") will receive the standard treatment and Kinesio tape lymphatic drainage technique application.
  The experimental group also receives the expected standard treatment, consisting in physiotherapeutic evaluation and physiotherapy counseling.
  Interventions: Device: Kinesio tape lymphatic drainage technique application
- Control group (No Intervention): Patients who belong to the control group ("CONTR") will receive only the standard treatment. Standard treatment consists in physiotherapy evaluation and counseling. The educational part, the demonstration of the exercises and the prosthesis mobilization are included in this treatment.

INTERVENTIONS:
Device: Kinesio tape lymphatic drainage technique application — Kinesio Tex Tape strips are applied following Dr.Kase draining techinique. The choice of tape's length and strips' number is based on the area of breast edema and/or presence of seroma, which must be completely covered. The patch is cut into fan strips. The major base is positioned near the functioning lymph node stations closest to the edema and/or seroma area. The bases and the tails of the fan must be applied with zero tension, while for the central part is reached 15-25% of tension. The first application takes place on the 1st post-operative day, while the second is performed on the 7th post-operative day. In case the tape is detached from one application to another, it is necessary that the patient resume in the clinic for a new application to ensure continuity of the therapeutic effect; otherwise the patient is eliminated from the study. The experimental group also receives the expected standard treatment, consisting in physiotherapeutic evaluation and counselin.
  Other Names: Kinesio Tape; Kinesiotape; Kinesio Tapes; Kinesio Taping; Kinesiology Taping
  Arms: Sperimental group

SUMMARY:
Over the last two decades in the field of oncology, the prevention, diagnosis, treatment and rehabilitation have reached a remarkable development, improving healing rates and reducing the number of deaths from cancer. The most frequent cancer in the female population is the breast one, which consequences can become disabling. In recent years, surgeons need to find more effective and less invasive treatments. Nowadays, despite the achievements, oncological surgery can cause side effects that cannot allow the return to normal life. Some of these problems are represented by the formation of edema and seroma, which can be handled by the physiotherapist through the manual lymphatic drainage and the application of an elastic tape. The elastic tape is used a lot in clinical practice, despite it lacks supportive evidence.

The primary aim of the study is to verify the effectiveness of Kinesio Tex Tape in reducing edema and seroma formation following complex reconstructive breast surgery. The secondary goals are the evaluation of the quality of the scar, of the perception of pain, of the degree of satisfaction and disability.

It is a controlled, monocentric, national, comparative, randomized, single-blind study. The sample size is 60 patients who undergo complex reconstructive breast surgery. Patients are divided into two groups: the experimental one (receiving standard treatment and Kinesio Tex Tape application) and a group of control (just receiving standard treatment). To evaluate edema and seroma, ultrasound is used; ultrasounds will be on the 1st, 15th and 30th postoperative days (T0, T1 and T2); Vancouver Scar Scale is used to define the quality of the scar (T0 and T2); to measure the subjective perception of pain and to evaluate the degree of patient satisfaction, two VAS scales are administered (the VAS scale for pain is administered at T0, T1 and T2, while the VAS scale for satisfaction is given at T1 and T2); Finally, to assess the degree of disability, the DASH Questionnaire is used (T0, T1 and T2).

DETAILED DESCRIPTION:
Screening at the first evaluation:

The anamnesis for each potentially eligible patient will be performed to assess whether the inclusion and exclusion criteria are met.

If the selection criteria for inclusion in the study are met, the patient will be proposed to participate in the study with the delivery of the patient information sheet and the form will be delivered to obtain written and signed informed consent.

Only after having signed the signature on the form, the patient will in fact be eligible for the study.

Randomization assigns to each patient the treatment strategy assigned by the random process, as well as the numerical code that uniquely identifies the patient in the study.

Once the randomization has been carried out, the following information will be collected at the moment before the tape application:

* Name and surname.
* Age.
* Profession.
* Type of surgical intervention.
* Side of the surgical intervention.
* Previous or concurrent diseases.
* Eventual adverse events.
* Thickness of skin and subcutaneous tissue, detected by ultrasound.
* Thickness of liquid, detected by ultrasound.
* Pain referred by the patient (VAS Scale).
* Patient satisfaction level (VAS Scale).
* Scar quality measured by the blind surgeon (Vancouver Scar Scale)
* Disability of the patient (DASH Questionnaire)

Screening for subsequent evaluations:

The following information will be collected:

* Thickness of skin and subcutaneous tissue (edema) and serum collection (seroma) detected by ultrasound.
* Quality of the scar measured by the blind surgeon (Vancouver Scar Scale).
* Subjective pain sensation (VAS Scale).
* Patient satisfaction level (VAS Scale).
* Disability of the patient (DASH Questionnaire).

Treatment:

Kinesio Tex Tape strips are applied to the patient in the experimental group following the technique of Dr. Kenzo Kase for lymphatic drainage. The choice of tape's length and of strips' number to be applied is based on the area of the breast edema and / or presence of seroma, which must be completely covered. The patch is cut into a fan strip: a length of kinesio tex tape is solid at one end and cut to create 4-6 narrow strips or tails. Corners are rounded to prevent detachment. The application area must be clean and dry. The major base is positioned near the functioning lymph node stations closest to the edema and / or seroma area. The bases and the tails of the fan must be applied with zero tension, while for the central part is reached 15-25% of tension, which is created manually or by extending the structures involved. Tails are applied in parallel, with a small distance between them.The first application takes place on the 1st post-operative day, while the second is performed on the 7th post-operative day. In the event that the tape is detached from one application to another, it is necessary that the patient resume in the clinic for a new application, so as to ensure continuity of the therapeutic effect; otherwise, the patient is eliminated from the study. The experimental group also receives the expected standard treatment. By standard treatment we mean physiotherapeutic evaluation and physiotherapy counseling. The educational part, the demonstration of the exercises to be performed autonomously and the demonstration of prosthesis mobilization are included in this treatment.

Temporary or ultimately treatment interruption:

There are no conditions that allows to interrupt and then restart the study. If a subject decides to interrupt the study, the decision will be ultimate and a conclusion visit will be carried out in order to understand the drop out motivations; data will be analysed for intention-to-treat analysis.

• Statistics considerations

Sample size:

In order to assess the 1st co-primary endpoint (seroma resolution at 30 days) the percentages will be compared; from our clinical experience we except the 50% of subjects without tape will resolve seroma at 30 days, while 90% of subjects with kinesio-tape treatment will resolve at the same time.

In order to highlight this difference we will need to recruit 30 subjects per group with 2,5 % alpha error and 80% statistical power.

Regarding the 2nd co-primary endpoint (edema reduction), taking as reference the mean of five ultrasound breast acquisition, a size of 30 subjects in each group and a 80% statistical power will be required to determine a difference of 1.69 mm between null hypothesis which establishes the mean of both groups is 10.00 mm and alternative hypothesis establishing the 2nd group mean is 8.31 mm, taking a standard deviation of 2.00 mm for both groups.

• Statistics analysis

Demographics data and outcomes in the study will be analysed through descriptive statistics.

In case of Gaussian distribution, the continuous variables will be described through mean and standard deviation, while in case non-Gaussian distribution the continuous variables will be described through median and interquartile range. Categorical variables will be described through frequency percentages.

Considered variables' normal distribution will be verified through Shapiro-Wilk Test.

For the 1st co-primary endpoint (seroma resolution) at 30 days proportions will be compared, and in order to make the survival analysis seroma resolution times will be considered.

Curves will be estimated through Kaplan and Meier method and two groups comparison will be carried out through log-rank test.

For the 2nd co-primary endpoint (edema reduction) means at 30 days will be compared through repeated measures analysis of variance.

The analysis will be conducted through intention-to-treat population analysis, considering the two groups as randomized.

Also a confirmation analysis will be conducted on population who has correctly carried out the treatment (per-protocol population).

• Ethical and regulating considerations:

This clinical study will be conducted according to the main laws drawn up by the 18th World Medical Assembly (Helsinki, 1964) and to all the applicable amendments drawn up by World Medical Assembly, and to the ICH guide lines for Good Clinical Practice.

This clinical trial will conducted with reference to all international laws and regulations, and to national laws and regulations in force in the Nation where it is carried out, as well as to each applicable guide line.

• Informed consent:

The investigator, or a person appointed by him and under his responsibility, will inform exhaustively participants about all aspects pertaining to the clinical trial, according to all the applicable regulating dispositions.

All participants will be exhaustively informed about the study, using words and language they will be able to understand.

Before taking part to the clinical trial the subjects will have had signed the informed consent forms.

The patients will be told they will be able to drop out the study whenever they want, without any requested explanations, and that their decisions will not have any consequence.

Every informed consent will be included in the investigator's files. The patient will be given a dated and signed copy of informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18;
* Complex reconstructive breast surgery with expander or prosthesis;
* Conditions favoring the correct execution of the proposed program (ability to complete the questionnaires);
* Written informed consent adherence.

Exclusion Criteria:

* Patients with psychic or other disorders that may prevent the completion of the questionnaires and / or informed consent adherence;
* Deferred breast reconstruction;
* Bilateral breast surgery reconstruction;
* Previous laterocervical emptying surgery;
* Maintenance of the surgical drainage for more than 8 days;
* Acute infections in other parts of the body.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-03 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in edema quantity at 30th postoperative day | The measurement is assessed at 1st, 15th and 30th post-operative days.
  Quantity of edema is measured in millimetres, through ultrasound scan. The verification of the effectiveness of elastic tape in terms of reduction of edema will be performed through ultrasound.
  During the ultrasound acquisition patients are indicated to assume the supine position on the couch, with 45 ° of humerus flexion and abduction, supported by an operator . Five points of maximum thickness of skin and subcutaneous tissue (edema) will be detected : retroareolar space, Upper-outer quadrant, Upper-inner quadrant, Lower-outer quadrant and Lower-inner quadrant. The thickness will be measured in millimeters.
Change in seroma quantity at 30th postoperative day | The measurement is assessed at 15th and 30th post-operative days.
  Quantity of seroma is measured in millimetres, through ultrasound scan. The verification of the effectiveness of elastic tape in terms of resolution of seroma will be performed through ultrasound.
  During the ultrasound acquisition patients are indicated to assume the supine position on the couch, with 45 ° of humerus flexion and abduction, supported by an operator . Five points of maximum thickness of liquid (seroma) will be detected : retroareolar space, Upper-outer quadrant, Upper-inner quadrant, Lower-outer quadrant and Lower-inner quadrant. The thickness will be measured in millimeters.

SECONDARY OUTCOMES:
Quality of the scar | The measurement is assessed at 1st and 30th post-operative days.
  The surgeon will make the evaluation of the quality of the scar using the Vancouver Scar Scale. The scale includes the following subscales: Pigmentation (M) in which the best score is "0 = normal" and the worst is "2= Hyperpigmented" , Pliability (P) in which the best score is "0 = normal" and the worst "5 = contracture", Height (H) in which the best score is " 0 = flat" and the worst is "3 = > 5 mm" and Vascularity (V) in which the best score is "0 = normal" and the worst is "3 = purple. The subscales' scores are summed to compute a total score, where lower values represent a better quality of the scar.
Subjective perception of pain | The measurement is assessed at 1st,15th and 30th post-operative days.
  The subjective perception of pain will be measured using Visual Analogue Scale for Pain. It is a measurement tool mainly used to indicate subjective pain characteristics. It consists of a strip of 10 cm in which its extremities correspond respectively to " 0 = no pain", "10 = worst pain that I can imagine", where lower values indicate a good subjective perception of pain. The health professional asks the patient to mark the pain perceived at that moment on the scale.
Degree of patient satisfaction | The measurement is assessed at 15th and 30th post-operative days.
  The degree of patient satisfaction will be measured using Visual Analogue Scale. It consists of a strip of 10 cm in which its extremities correspond respectively to "0 = no satisfaction", "10 = maximum satisfaction", where higher values indicate a good degree of satisfaction. The health professional asks the patient to mark the satisfaction perceived at that moment on the scale.
Degree of disability | The measurement is assessed at 1st, 15th and 30th post-operative days.
  The degree of disability will be measured using DASH scale (The Disability of the Arm, Shoulder and Hand). It is a questionnaire concerning symptoms and abilities to perform certain activities that mainly require the use of the upper limb. For each subscale (30 items) the best score is "1 = no difficulty" and the worst is "5 = unable". The patient is asked to assign a score from 1 to 5 for each activity reported by referring only to the operated side. For the activities contraindicated by the surgeon patients are suggested to give score 5, "unable".
  On the 15th and 30th post-operative day the questions related to the activities of daily life refer to the past week, while on the 1st post-operative day the patients are required to consider the time passed since the intervention. The subscales' scores are summed to compute a total score, where lower values represent a lower degree of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Martella, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCSSRaffaele, Milan, Italy